CLINICAL TRIAL: NCT02133534
Title: The Effect of Atorvastatin on Endothelial Cell Dysfunction in Chronic Kidney Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: failure to enroll
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00011172
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Kidney Disease; High Cholesterol
Keywords: Chronic kidney disease; High cholesterol
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypercholesterolemia | interventions — Atorvastatin

ARMS (1):
- Atorvastatin (Experimental): Subjects will be treated with atorvastatin 10 mg/day for 30 days. The study team will obtain one blood and urine sample at baseline prior to starting atorvastatin therapy, and again after 30 days of drug therapy. The study team will do ultrasound imaging of the arm in which a probe will be placed over the blood vessels to measure the diameter of the artery and how this changes after a blood pressure cuff is inflated and then deflated. Subjects will take one nitroglycerine tablet during the ultrasound imaging.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin
  Other Names: Lipitor

SUMMARY:
The purpose of this study is to see if patients with chronic kidney disease have endothelial cells that don't function properly, which is thought to be a marker for cardiovascular risk. Endothelial cells line the heart and blood vessels. The investigators will treat your high cholesterol with a cholesterol-lowering drug (atorvastatin, or Lipitor). They will determine if this cholesterol lowering drug improves subjects' cholesterol as well as the function of endothelial cells.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3, 4 and 5 chronic kidney disease (not on dialysis)
* Hyperlipidemia requiring cholesterol lowering therapy
* Aged 18 to 80 years old
* Ability to provide informed consent

Exclusion Criteria:

* Patients requiring multiple cholesterol reducing agents
* Patients with neovascularization present, such as neoplasm, active wounds, or significant retinopathy
* Patients with contraindications or allergy to statins

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Szczech, MD, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin: Subjects will be treated with atorvastatin 10 mg/day for 30 days. The study team will obtain one blood and urine sample at baseline prior to starting atorvastatin therapy, and again after 30 days of drug therapy. The study team will do ultrasound imaging of the arm in which a probe will be placed over the blood vessels to measure the diameter of the artery and how this changes after a blood pressure cuff is inflated and then deflated. Subjects will take one nitroglycerine tablet during the ultrasound imaging.
  Atorvastatin
Period: Overall Study
Arm/Group | Atorvastatin
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Atorvastatin
Number analyzed (Participants) | 1
Age, Customized [Number; unit: participants]
  Greater than 18 Years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Improved Counts of Endothelial Progenitor Cells
Description: Improvement of endothelial cell (EC) dysfunction will be assessed by improved counts of endothelial progenitor cells.
Time Frame: baseline, 30 days
Population: Early termination because of insufficient accrual. With only one study participant, data could not be analyzed.
Arm/Group | Atorvastatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: Early termination because of insufficient accrual. With only one study participant, data could not be analyzed.
Arm/Group | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Early termination of trial due to lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No